CLINICAL TRIAL: NCT04373382
Title: Peer Champion Support for Hospital Staff During and After the COVID-19 Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Robert Maunder, Professor, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 20-0084-E
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Burnout
Keywords: healthcare workers; resilience; infectious disease; COVID-19; burnout
MeSH Terms: conditions — Burnout, Psychological; Communicable Diseases; COVID-19

STUDY DESIGN:
Intervention Model Description: Hospital staff will receive support from Peer Resilience Champions, whose activities will, in part, be modelled on the role that psychiatrists acting as support coaches have played in during the acute phase of the pandemic. These include support, identification of needs, education, advocacy and resource navigation. In doing so, they follow evidence-based principles and guidelines.
  A randomized cluster stepped wedge design will be used, with five clusters of clinical units and departments constructed in order to approximate the following goals: similar number of staff, comparable COVID-19 exposure, similar mix of staff by discipline and gender, number of clusters small enough to allow for the PRC intervention to be provided with at least six months of implementation within the two-year study after cross-over occurs. (Two arms).
  The Enriched survey intervention will be a randomized controlled trial design with equal allocation (1:1) to both the express and enriched surveys. (Two arms).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Peer Resilience Champion Support (Experimental): The clusters that receive this intervention will receive support from a Peer Resilience Champion.
  Interventions: Behavioral: Peer Resilience Champion
- No Peer Resilience Champion Support (No Intervention): The clusters in this arm of the study will not receive the Peer Resilience Champion support until they cross-over into the Peer Resilience Champion support arm.
- Enriched Feedback (Experimental): This arm of the study encompasses individuals who will receive feedback from the survey that will hopefully help provoke self-reflection.
  Interventions: Behavioral: Enriched Survey Feedback
- Express Feedback (No Intervention): This arm of the study encompasses individuals who will not receive feedback from the survey.

INTERVENTIONS:
Behavioral: Peer Resilience Champion — PRC is supplied to everyone and provides support to hospital staff during the COVID-19 pandemic in a stepped-wedge design.
  Arms: Peer Resilience Champion Support
Behavioral: Enriched Survey Feedback — This intervention provides feedback based on answers to questionnaires to those in the Enriched Feedback arm of the study.
  Arms: Enriched Feedback

SUMMARY:
Experience from the 2003 Severe Acute Respiratory Syndrome (SARS) outbreak taught that healthcare workers (HCWs) often experience chronic stress effects for months or years after such an event, and that supporting HCWs requires attention to the marathon of occupational stress, not just the sprint of dramatic stressors that occur while infections are dominating the news. This study will test if the well-being of hospital workers facing a novel coronavirus outbreak is improved by adding either of two interventions: (1) Peer Resilience Champions (PRC): an interdisciplinary team of professionals who actively monitor for early signs of heightened stress within clinical teams, liaise between staff and senior management to improve organizational responsiveness, and provide direct support and teaching (under the supervision of experts in resilience, infection control, and professional education). Investigators will test the effectiveness of this PRC Intervention by rolling it out to different parts of the hospital in stages and comparing levels of burnout before and after the intervention reaches particular teams and units (a stepped wedge design). By the end of the study, PRC Support will have been provided to all clinical and research staff and many learners (> 6,000 people). Note that the provision of PRC support will be directed to the entire organization. The research portion of the study is the evaluation of PRC support through a repeated survey completed by consenting staff. Investigators will test the effectiveness of the PRC by measuring trends in burnout and other effects of stress over the course of the study in a subgroup of hospital workers (as many as consent, target ~1000 people) through an online questionnaire (called "How Are You?"). (2) The second intervention is an enriched version of the "How Are You?" Survey, which provides personalized feedback about coping, interpersonal interactions and moral distress. Participants will be randomized (1:1) to receive the shorter Express Survey (identifying data and outcome measures only), or the Enriched survey (all of the Express measures plus additional measures with feedback based on responses). It is hypothesized that both the PRC intervention and the Enriched Survey intervention will help prevent or reduce instances of burnout in HCWs.

DETAILED DESCRIPTION:
This project studies the impact of two interventions, the addition of Peer Resilience Champions to other hospital supports and an interactive computer-based learning intervention that provides personalized feedback about relevant interpersonal and psychological characteristics of participants.

The Peer Resilience Champion (PRC) Intervention Investigators will second or hire an interdisciplinary team of healthcare professionals (e.g. nurses, social worker, or infection control professional, total of 1 FTE) to serve as Peer Resilience Champions. These Champions will receive coaching and then ongoing supervision in the relevant aspects of stress management, peer support, and resource navigation by expert members of the research team based on existing evidence. Peer Resilience Champions will act predominantly at the level of clinical units and departments.

The activities of Peer Resilience Champions will, in part, be modelled on the role that psychiatrists acting as support coaches have played in during the acute phase of the pandemic. These include support, identification of needs, education, advocacy and resource navigation. In doing so, the Champions follow evidence-based principles and guidelines. The model is to provide quickly responsive, adaptive, peer support because it is expected that the needs of staff will change over the course of a pandemic and in its aftermath.

Peer Resilience Champions will work in an expanding selection of hospital locations, following a randomized cluster (stepped wedge) design until the resource is available to the entire organization. People who work and learn at Sinai Health do not need to participate in this study in order to receive the potential benefits provided by Peer Resilience Champions, which will be provided irrespective of study participation. The effectiveness of Peer Resilience Champions in reducing burnout and other outcomes will be tested using outcome measures included in the feedback staff survey (see below), which is completed by consenting participants in this study.

Interactive Computer-based Learning Intervention A staff survey which includes all primary and secondary outcomes measures will be completed by consenting participants at intervals of approximately 3 months seven times (over approximately 21 months). Participating staff will be randomized 1:1 to receive only these measures with no feedback (the Express Survey) or these measures plus additional measures of interpersonal and psychological characteristics, with personalized feedback (the Enriched Survey). Feedback is based on previous experience from the investigators in providing feedback from validated measures completed online to both healthcare workers and the general public. The purpose of feedback is to encourage self-reflection, especially with respect to coping and interpersonal interactions. The core measures that are common to both the Express and Enriched surveys serve to tests the effectiveness of the Peer Resilience Champions Intervention. The effectiveness of the Interactive Computer-based learning intervention will be tested by comparing the core measures between those receiving the Express Survey and those receiving the Enriched Survey.

Peer Resilience Champion Support The study design provides a controlled comparison of support as usual to PRC support. Using a randomized cluster (stepped wedged) design, usual staff support will be compared to that of PRC. PRC operates largely at the level of the clinical units and groups, and so a randomized cluster design is preferable to a randomized controlled trial. The stepped wedge design allows clusters of hospital staff/volunteers to receive the PRC intervention in a random sequence until the resource is available to all areas of the hospital.

This intervention will take place at Sinai Health System, including the Mount Sinai (approximately 4500 employees), Bridgepoint (approximately 1200 staff), and Lunenfeld-Tanenbaum Research Institute (LTRI) (approximately 1200 staff).

Five clusters of clinical units and departments will be constructed that are approximately balanced between hospital units and staff groups with (i) high COVID patient acuity (ICU, Emergency, medical units with negative pressure rooms) or high exposure to patients from community with unknown COVID status (Family Medicine, Labour and Delivery), (ii) all other clinical patient care areas, (iii) non-patient care areas, and (iv) areas in which most or all staff are/were temporarily restricted from attending the hospital (e.g. LTRI, volunteers).

After survey participants (and their disciplines and clinical units) are identified (T0 survey), their corresponding units, will be grouped into one of the five clusters in order to meet the above goals. These clusters will then be randomized in order to determine the order of intervention implementation. Each cluster will either receive support as usual or PRC for a period of three months, followed by the completion of a survey questionnaire given at seven different time points (T1-T7) spaced by three months.

NOTE - justification for choosing a non-blind comparison: Since the Express Survey is shorter than the Enriched Survey, participants are not blind to survey cohort assignment. Nor does the design control for time spent on an online activity. It would be possible to control for the duration of the survey by expanding the length of the control condition and this would also allow for the possibility of a blind comparison. However, a longer control survey would increase the risk of drop-out among participants in the control condition because completing surveys without interaction or feedback is not interesting. Since maximizing continued participation in serial surveys is critical to testing the PRC intervention hypothesis, a non-blind test of the Enriched Survey intervention hypothesis is preferable to increasing the risk of being underpowered to test the PRC hypothesis.

Feedback Surveys Immediately after consenting, participants will be asked to complete the T0 survey that asks about identifying information, and the characteristics of the participant's work at Sinai Health. The T0 survey also collects an email address, to which all subsequent surveys (T1 to T7) are sent. Following receipt of the T0 survey, participants are randomized to receive either the Express Survey (T1 to T7) or the Enriched survey (T1 to T7). In either case, T1 is sent soon (~1-2 weeks) after T0. All subsequent surveys are sent at approximately 3-month intervals.

T0 survey - The initial survey collects identifying data (non-binary gender, discipline, department, age, marital status), years of experience, SARS experience, number of people in household and information about COVID-19 experience to date (exposure to patients, experience with isolation of self or family members, testing etc.). Two free optional text write-in questions provide allow participants to describe more about themselves or their experience (past experience surveying healthcare workers post-SARS was that many were keen to write at length about their experience, beyond data collected more formally, and that insights from this open-ended reporting were valuable for placing quantitative results in experiential context during analysis and knowledge dissemination phases). The T0 survey takes about 10 minutes to complete plus whatever time is spent providing optional free-text answers.

Express Survey: The express survey includes validated measures of the primary outcome, the emotional exhaustion scale of the Maslach Burnout Inventory. The Express Survey also includes measures of secondary outcomes: sleep, post-traumatic stress disorder symptoms, psychological distress, occupational resilience, and COVID-19 prevention and control self-efficacy (using an instrument revised from a measure of self-efficacy used in preparation for an expected pandemic. The survey is the same each time it is completed (T1 to T7) at 3-month intervals. The Express Survey takes about 10 minutes to complete.

Enriched Survey: The Enriched Survey contains all of the measures included in the Express survey. No feedback is provided from any of these measures (i.e. this portion of the Enriched survey is identical to the Express Survey). In addition to these core outcome measures, the Enriched Survey includes measures of personality, interpersonal style and coping and provides personalized feedback based on scores at time points T1 to T6. The interactive measures included vary from one survey time point to the next in order to provide variety, and to cover a larger number of participant characteristics within the limits of reasonable survey time burden. State-dependent characteristics which may change over time (coping, interpersonal problems) are measured twice. A measure of lifetime experience with moral distress and a measurement of attachment, a stable trait, occur only once. The Enriched T1 to T6 surveys take about 10-20 minutes.

Sample size This study is powered to test hypothesis 1, which is expected to require a larger sample size than testing hypothesis 2. There are over 6000 staff at Sinai Health. Assuming a starting proportion of 30.4% of staff with high burnout (based on previous studies), an 80% power, and an alpha level of 0.05, five clusters of 200 staff providing measures per cluster is sufficient to detect a drop of ≥ 9.4% (with an intracluster correlation coefficient [ICC] of 0.01), ≥10.7% (ICC of 0.015), or ≥ 11.9% (ICC of 0.2). These ICC estimates are congruent with previous studies. These differences are consistent with a post-SARS study that found high burnout in 30.4% of exposed and 19.2% of unexposed HCWs. Five clusters of 200 staff (n=1000) would require <17% of staff to consent to participate and complete the measures.

ELIGIBILITY:
Inclusion Criteria:

* An employee, physician, scientist, employee of a contractor or retail business, learning, or volunteer of Sinai Health at time of recruitment. Must be able to read and respond to a survey in English. Need to have access to a computer or device connected to the internet and be able to use said device.

Exclusion Criteria:

* Failure to meet inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 882 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2023-07-27 (Estimated)

PRIMARY OUTCOMES:
Change in instances of burnout for hospital staff due to the Peer Resilience Champion intervention | 21 months
  Impact of the Peer Resilience Champion intervention as determined by a high outcome (defined as a cutoff of ≥27 on the Maslach Burnout Inventory: Emotional Exhaustion subscale)
Change in instances of burnout for hospital staff due to the Enriched Feedback Survey intervention | 21 months
  Impact of the Enriched survey feedback intervention as determined by a high outcome (defined as a cutoff of ≥27 on the Maslach Burnout Inventory: Emotional Exhaustion subscale)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Maunder, Principal Investigator — Sinai Health
Locations (1):
- Sinai Health System, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maunder RG, Lancee WJ, Balderson KE, Bennett JP, Borgundvaag B, Evans S, Fernandes CM, Goldbloom DS, Gupta M, Hunter JJ, McGillis Hall L, Nagle LM, Pain C, Peczeniuk SS, Raymond G, Read N, Rourke SB, Steinberg RJ, Stewart TE, VanDeVelde-Coke S, Veldhorst GG, Wasylenki DA. Long-term psychological and occupational effects of providing hospital healthcare during SARS outbreak. Emerg Infect Dis. 2006 Dec;12(12):1924-32. doi: 10.3201/eid1212.060584. PMID 17326946
- [Background] Maunder R. The experience of the 2003 SARS outbreak as a traumatic stress among frontline healthcare workers in Toronto: lessons learned. Philos Trans R Soc Lond B Biol Sci. 2004 Jul 29;359(1447):1117-25. doi: 10.1098/rstb.2004.1483. PMID 15306398
- [Background] Salyers MP, Bonfils KA, Luther L, Firmin RL, White DA, Adams EL, Rollins AL. The Relationship Between Professional Burnout and Quality and Safety in Healthcare: A Meta-Analysis. J Gen Intern Med. 2017 Apr;32(4):475-482. doi: 10.1007/s11606-016-3886-9. Epub 2016 Oct 26. PMID 27785668
- [Background] Edmondson AC, Higgins M, Singer S & Weiner J. Understanding Psychological Safety in Health Care and Education Organizations: A Comparative Perspective. Research in Human Development. 2016; 13(1): 65-83.
- [Background] Maunder RG, Lancee WJ, Mae R, Vincent L, Peladeau N, Beduz MA, Hunter JJ, Leszcz M. Computer-assisted resilience training to prepare healthcare workers for pandemic influenza: a randomized trial of the optimal dose of training. BMC Health Serv Res. 2010 Mar 22;10:72. doi: 10.1186/1472-6963-10-72. PMID 20307302
- [Background] Aiello A, Khayeri MY, Raja S, Peladeau N, Romano D, Leszcz M, Maunder RG, Rose M, Adam MA, Pain C, Moore A, Savage D, Schulman RB. Resilience training for hospital workers in anticipation of an influenza pandemic. J Contin Educ Health Prof. 2011 Winter;31(1):15-20. doi: 10.1002/chp.20096. PMID 21425355